CLINICAL TRIAL: NCT00762125
Title: Subgroups of Fibromyalgia Syndrome (FMS): Symptoms, Beliefs, and Tailored Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Dennis Turk, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AR044724-07 (NIH); R01AR044724-07 (NIH)
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia Syndrome; FMS; Physical Therapy; Psychotherapy; Group Counseling; Individual Counseling; Chronic Pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- Cognitive restructuring and coping skills training (CR+ST) (Experimental)
  Interventions: Behavioral: CR+ST
- Exposure therapy (ET) (Experimental)
  Interventions: Behavioral: ET
- Combination (COMB) treatment (Experimental)
  Interventions: Behavioral: CR+ST; Behavioral: ET
- Attention control (AC) treatment (Active Comparator)
  Interventions: Behavioral: AC treatment

INTERVENTIONS:
Behavioral: CR+ST — Addresses maladaptive beliefs in general and includes education and training in the use of specific coping strategies
  Arms: Cognitive restructuring and coping skills training (CR+ST); Combination (COMB) treatment
Behavioral: ET — Addresses beliefs and emotional arousal during confrontations with feared element (exercising) through use of counter-conditioning and corrective feedback
  Arms: Combination (COMB) treatment; Exposure therapy (ET)
Behavioral: AC treatment — Provides support and controls for nonspecific factors associated with exposure to therapists and other FMS sufferers, but does not directly address either maladaptive beliefs or emotional arousal
  Arms: Attention control (AC) treatment

SUMMARY:
Fibromyalgia syndrome (FMS) refers to a set of symptoms that include exhaustion, muscle pain, and tender points, where slight pressure can cause pain. Doctors do not know what causes FMS or how to cure it, but some treatments have helped relieve its symptoms. Progressive exercise, in which exercise is started at low levels and then increased, is one of the most reliable treatments, but people with FMS often avoid exercise or stop after completing exercise programs. This research will focus on the idea that people with FMS do not exercise because they are afraid of injury or have had a negative experience exercising. Participants will undergo one or a combination of several different treatments that aim to reduce fear of exercising. The different treatments will then be evaluated on their effectiveness in reducing disability among people with FMS.

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) is a condition without a known cause or cure. Differing theories place the blame on abnormal sensitivity to pain receptors in the brain, changes in metabolism and hormones, abnormalities in the autonomic nervous system, sleep disturbances, infection, or injury. A diagnosis of FMS, therefore, is based on a set of symptoms. These include pain in muscles, ligaments, and tendons; fatigue; and multiple tender points on the body, where even slight pressure causes pain.

Although there is no cure, FMS can be treated to reduce the severity or presence of symptoms. One of the most reliable ways to do this is through progressive exercise, which involves starting at low levels of exercise and building up to longer and more strenuous levels. Despite the benefit of exercise, FSM sufferers often drop out of supervised exercise programs or discontinue exercise once they are no longer supervised. Some FMS patients may have a fear-based avoidance of exercise, believing it will provoke pain or deterioration of their condition and experiencing significant negative emotional arousal when they exercise. This may be due to a prior painful or uncomfortable experience while exercising.

This study will employ multiple treatments that are usually used for treatment of phobias and will aim to reduce fear, increase exercising, and improve FMS symptoms. Under the purview of cognitive behavioral therapy (CBT) are multiple types of treatments. Cognitive restructuring (CR) and coping skills training (ST) paired together address maladaptive beliefs and facilitate the development of more effective coping strategies. Exposure therapy (ET) reduces the level of emotional arousal when patients are exposed to the feared stimulus, in this case exercising. Attention control (AC) treatment, not a type of CBT, provides patients with support and controls for nonspecific factors related to exposure to their feared stimulus. AC will be used as the control treatment in this study.

Participation in this study will last 4 months. After recruitment and an initial evaluation, participants will be placed on a waiting list for 8 weeks to determine whether their symptoms improve or change naturally. They will then be reassessed and randomly assigned to one of the following groups for 8 weeks of treatment:

1. CR+ST: This group will help participants develop adaptive ways of thinking and acting to alter maladaptive beliefs in general and beliefs about certain exercises in specific.
2. ET: This group will help participants to decrease their fear response during specific exercises through progressive, controlled exposure to the feared stimulus.
3. COMB: This group will combine CR+ST and ET treatment plans so that adaptive thoughts and behaviors will be emphasized in the first 4 weeks, and exposure to feared stimuli will be emphasized in the second 4 weeks.
4. AC: This group will offer participants non-directive, supportive counseling. Each treatment group will meet in weekly 90-minute group sessions for the first 4 weeks and in weekly 60-minute individual sessions for the second 4 weeks. Participants will have 60-minute physical therapy sessions accompanying every treatment session. Participants will also be given weekly homework assignments specific to their treatment group.

Participants will undergo a series of assessments that include self-report measures, medical and psychological evaluations, and a physical capability evaluation by a physical trainer. These assessments will be performed at recruitment, after the 8-week waiting period, after treatment, at 1- and 3-month mail and telephone follow-ups, and at a 6-month follow-up in the treatment clinic. They will assess fear, health, physical ability, and psychological health.

ELIGIBILITY:
Inclusion Criteria:

* Meet American College of Rheumatology (ACR) criteria for the diagnosis of fibromyalgia
* Able to comply with functional assessment and treadmill exercise

Exclusion Criteria:

* History of psychiatric hospitalization, suicide attempt, or significant problems with chemical dependency during the 6 months prior to enrollment in the study
* Evidence of severe psychiatric disorder that would prevent participation
* Medical conditions, such as significant cardiac disease, that make it medically unsuitable for participation in a progressive exercise program
* A medical condition, such as multiple sclerosis, that has a high likelihood of obscuring effects of the experimental treatments
* Anxiety or mood disorders in which symptoms are severe enough to prevent participation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2005-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | Measured at the initial evaluation; after 8 weeks on a waiting list; immediately after treatment; and 1, 3, and 6 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Dennis C. Turk, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States